CLINICAL TRIAL: NCT03935555
Title: Phase 1b Study of PU-H71 for the Treatment of Subjects With Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (Post-PV MF), Post-Essential Thrombocythemia Myelofibrosis (Post-ET MF), Treated With Ruxolitinib
Brief Title: Assess the Safety, Tolerability Oral PU-H71 in Subjects Taking Ruxolitinib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Samus Therapeutics company closure
Sponsor: Samus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PU-H71-01-003
Record Dates: First submitted 2019-03-14; First posted 2019-05-02 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Primary Myelofibrosis (PMF); Post-Polycythemia Vera Myelofibrosis (Post-PV MF); Post-Essential Thrombocythemia Myelofibrosis (Post-ET MF)
Keywords: Primary Myelofibrosis (PMF); Post-Polycythemia Vera Myelofibrosis (Post-PV MF); Post-Essential Thrombocythemia Myelofibrosis (Post-ET MF)
MeSH Terms: conditions — Primary Myelofibrosis | interventions — 9H-purine-9-propanamine, 6-amino-8-((6-iodo-1,3-benzodioxol-5-yl)thio)-N-(1-methylethyl)-

STUDY DESIGN:
Intervention Model Description: The study will employ a standard 3+3 dose escalation design to determine maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D), with additional subjects treated in a dose expansion cohort. The time period for collecting dose limiting toxicities (DLTs) is 1 cycle (21 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Oral - 50mg (Experimental): PU-H71 (a small molecule purine-scaffold epichaperome inhibitor selective for stress-induced HSP90 in epichaperomes).
  Interventions: Drug: PU-H71
- Oral -100 mg (Experimental): PU-H71 (a small molecule purine-scaffold epichaperome inhibitor selective for stress-induced HSP90 in epichaperomes).
  Interventions: Drug: PU-H71
- Oral - 200 mg (Experimental): PU-H71 (a small molecule purine-scaffold epichaperome inhibitor selective for stress-induced HSP90 in epichaperomes).
  Interventions: Drug: PU-H71
- Oral - 300 mg (Experimental): PU-H71 (a small molecule purine-scaffold epichaperome inhibitor selective for stress-induced HSP90 in epichaperomes).
  Interventions: Drug: PU-H71

INTERVENTIONS:
Drug: PU-H71 — PU-H71 is a synthetic purine-scaffold stress chaperome inhibitor, which specifically targets HSP90 in the tumor-specific epichaperome

SUMMARY:
This is a multicenter, Phase 1b study with dose escalation and expansion cohorts designed to assess the safety, tolerability, PK, and preliminary efficacy of PU-H71 in subjects with PMF, Post-PV MF, Post-ET MF, taking stable doses of ruxolitinib.

DETAILED DESCRIPTION:
The study will employ a standard 3+3 dose escalation design to determine maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D), with additional subjects treated in a dose expansion cohort. The time period for collecting dose limiting toxicities (DLTs) is 1 cycle (21 days).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide written informed consent before any study-specific procedures are performed.
2. Subject is willing to comply with all study procedures and restrictions.
3. Subject is ≥18 years of age.
4. Subject has confirmed diagnosis of PMF, Post-PV MF, or Post-ET MF.
5. Subject has been receiving ruxolitinib therapy meeting the following criteria:

   * Receiving ruxolitinib >3 months prior to enrollment.
   * Stable dose for 8 weeks before starting therapy with PU-H71.
6. Subject with evidence of evaluable residual burden of disease following ruxolitinib monotherapy treatment, consisting of:

   • Persistent or worsening disease-related symptoms, including but not limited to fatigue, pruritus, night sweats, early satiety, and other symptoms as determined by a Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) score of >12 points.

   AND

   • Documented splenomegaly of at least 5 cm below the costal margin as measured on inspiration by physical examination.
7. Subject has an Eastern Cooperative Oncology Group performance status of 0 to 2.
8. Acceptable pre-study organ function during screening defined as:

   * Absolute neutrophil count (ANC) ≥1000/µL.
   * Platelet count ≥50,000/µL.
   * Alanine aminotransferase or aspartate aminotransferase ≤2×upper limit of normal.
   * Direct serum bilirubin ≤ 1.5×upper limit of normal.
   * Creatinine clearance >50 mL/min/1.73 m2 based on the Cockcroft Gault equation.
9. If female and of childbearing potential (premenopausal and not surgically sterile), the subject:

   * Must have a negative serum or urine pregnancy test at screening. The serum pregnancy test must be obtained prior to the first administration of PU-H71 (≤72 hours prior to dosing) in all premenopausal women and women <2 years after the onset of menopause.
   * Must agree to use an acceptable method of effective contraception for the duration of the study and for 13 weeks after receiving the last dose of study treatment.
10. If male, the subject agrees to:

    * Use an acceptable method of effective contraception for the duration of the study and for 13 weeks after receiving study treatment.
    * Agrees to abstain from sperm donation for the duration of the study and for 13 weeks after receiving the last dose of study treatment

Exclusion Criteria:

1. Subject has known active liver disease, including viral hepatitis or cirrhosis.
2. Subject has known or suspected human immunodeficiency virus (HIV) or other active infections requiring acute or chronic treatment with systemic antibiotics. Conditions requiring topical antibiotics are acceptable.
3. Subject has a QT interval corrected using Fridericia's formula (QTcF) >480 ms (corrected) in the screening or baseline ECG based on median value of ECG's obtained.
4. Subject has left ventricular ejection fraction (LVEF) ≤50%, or below institution's lower limit of normal (whichever is lower), by echocardiogram or multigated acquisition (MUGA) scan.
5. Subject has a history (or family history) of long QT syndrome.
6. Subject has coronary artery disease with an ischemic event within 6 months prior to screening.
7. Subject has a permanent cardiac pacemaker.
8. Subject has history of a second primary malignancy within the past 2 years, except for the following (if appropriately treated and considered cured): Stage I endometrial, surgically treated cervical or prostate carcinoma, and non-melanoma skin cancer.
9. Subject has significant uncontrolled medical condition within 6 months prior to screening, as determined by the Investigator.
10. Subject has planned use of antineoplastic agents (chemotherapy or cytotoxic drugs), immunotherapy, experimental therapy, or biologic therapy for treatment of MPN with the exception of ruxolitinib.
11. Subject uses systemic corticosteroids (ie, prednisone >12.5 mg/day or dexamethasone >2 mg/day) within 2 weeks prior to Cycle 1 Day 1.
12. Subject has planned or current use of strong CYP3A4/5, CYP2D6, or CYP2C19 inhibitors or inducers within 1 week or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
13. Subject has planned or current use of medications that carry a risk for Torsades de Pointes within 1 week or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
14. Subject has planned or current use of herbal preparations/medications at least 7 days prior to Cycle 1 Day 1.
15. Subject has previously received PU-H71.
16. Subject has concurrent participation in any interventional studies (except PU-H71-Positive Emission Tomography (PET) Scan Studies) within 14 days or 5 half-lives (whichever duration is longer) of Cycle 1 Day 1.
17. Subject has uncontrolled diabetes mellitus, in the judgment of the Investigator.
18. Subject has any other condition or laboratory abnormality or receives any other treatment(s) that may increase the risk associated with study participation or may interfere with the interpretation of study results in the judgment of the Investigator.
19. Subject has an active ocular condition that in the opinion of the Investigator, may alter visual acuity during the course of the study (ie, ocular inflammatory disease, etc.) or a history or anticipation of major ocular surgery (including cataract extraction, intraocular surgery, etc.) during the study.
20. Women who are pregnant or breastfeeding or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Assess Safety, Tolerability and Pharmacokinetics of PU-H71 | 24 weeks
  Determine the human exposure PK including Cmax
Assess Safety, Tolerability and Pharmacokinetics of PU-H71 | 24 weeks
  Determine the human exposure PK including Tmax
Assess Safety, Tolerability and Pharmacokinetics of PU-H71 | 24 weeks
  Determine the human exposure PK including AUC0-t
Assess Safety, Tolerability and Pharmacokinetics of PU-H71 | 24 weeks
  Determine the human exposure PK including AUC0-inf
Assess Safety, Tolerability and Pharmacokinetics of PU-H71 | 24 weeks
  Determine the human exposure PK including CL
Assess Safety, Tolerability and Pharmacokinetics of PU-H71 | 24 weeks
  Determine the human exposure PK including t1/2
Assess Safety and Tolerability of PU-H71 | 24 weeks
  Determine the Incidence and severity of AEs as determined by the NCI-CTCAE Version 5.0 and by changes in physical examinations
Assess Safety and Tolerability of PU-H71 | 24 weeks
  Determine the Incidence and severity of AEs as determined by the NCI-CTCAE Version 5.0 and by changes in electrocardiograms (ECGs)
Assess Safety and Tolerability of PU-H71 | 24 weeks
  Determine the Incidence and severity of AEs as determined by the NCI-CTCAE Version 5.0 and by changes in vital signs
Assess Safety and Tolerability of PU-H71 | 24 weeks
  Determine the Incidence and severity of AEs as determined by the NCI-CTCAE Version 5.0 and by changes in clinical laboratory evaluations
Assess treatment response of PU H71 | 24 weeks
  Treatment response in myelofibrosis (MF) is to be evaluated using the revised International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT)
Assess treatment response of PU H71 | 24 weeks
  Treatment response in myelofibrosis (MF) is to be evaluated using the revised European LeukemiaNet (ELN) response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverman, M.D., Study Director — Samus Therapeutics
Locations (3):
- United States (3):
  - Marin Cancer Care - Greenbrae (California Cancer Care A Medical Group, Inc. - Greenbrae), Larkspur, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No